CLINICAL TRIAL: NCT05673941
Title: "InMotion" - Physical Training With Creative Movement as an Intervention for Adults With Schizophrenia
Acronym: InMotion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 278241
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Schizophrenia; Physical activity; Randomized trial; EEG; fNIRS; Motion capture; Dance; Creative movement; Physical Training
MeSH Terms: conditions — Schizophrenia; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be pseudonymized by using a study code. The researchers will be blind to group allocation when analyzing data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative movement (Experimental): The intervention will be performed as a group activity twice a week during a 12-week period. Each group will include 4-6 participants under the guidance of two instructors, and a related party if needed or wanted from the participant. The exercise is partly accompanied with calm music and recorded nature sounds and partly made in silence listening to one's own bodily rhythm. The exercise consists of tasks related to cardio and strength training, balance, conscious breathing, body awareness, mental imagery (nature visualizations), flexibility, emotional expression, and movement anticipation together with the facilitator and fellow participants. All the tasks are practiced during a flow of 45- to 60-minute exercise without any major breaks. Complexity and physical intensity of the tasks will gradually increase over the 12-week intervention period.
  Interventions: Other: Creative physical training
- Control group (No Intervention): The control group receives standard medical care and gets access to the intervention in digital form after the study has ended.

INTERVENTIONS:
Other: Creative physical training — The intervention will be performed as a group activity twice a week during a 12-week period. Each group will include 4-6 participants under the guidance of two instructors, and a related party if needed or wanted from the participant. The exercise is partly accompanied with calm music and recorded nature sounds and partly made in silence listening to one's own bodily rhythm. The exercise consists of tasks related to cardio and strength training, balance, conscious breathing, body awareness, mental imagery (nature visualizations), flexibility, emotional expression, and movement anticipation together with the facilitator and fellow participants. All the tasks are practiced during a flow of 45- to 60-minute exercise without any major breaks. Complexity and physical intensity of the tasks will gradually increase over the 12-week intervention period.
  Arms: Creative movement

SUMMARY:
InMotion is a randomized controlled study where adults with schizophrenia and schizophrenia-similar conditions, will be recruited to receive physical training with creative movements as an intervention, twice a week for a period of 12 weeks. The main outcome is changes in schizophrenia-related symptoms, secondary outcomes are changes in quality of life, physical and cognitive function, brain activity, and how the intervention is experienced by the participants.

DETAILED DESCRIPTION:
Schizophrenia (SCZ) is among the world's top ten causes of long-term disability (World Health Organization, 2004). The major symptoms of SCZ include hallucinations, delusions, affective flattening, apathy and cognitive impairment. These symptoms lead to major problems in social and occupational functioning, and in self-care.

Our primary aim is to investigate the effects of 12-weeks of physical training with creative movement as an intervention given in addition to ongoing pharmacological treatment, in treating SCZ-symptoms compared to a control group. Secondary aim is to provide results regarding the effects of the intervention on (a) clinical symptom measures and quality of life, (b) levels of physical activity, physical function and measures of general health indicators, (a) clinical symptom measures and quality of life, (b) levels of physical activity, physical function and measures of general health indicators, (c) error detection and conflict resolution on the prefrontal cortex, memory and context processing (d) fluency of speak, and (e) emotional induction and regulation on specific emotions on the frontal cortex. Trough qualitative interviews, we will examine the participants' and their relative parties' experiences from taking part of the intervention and eventual experienced effects from it.

This study, called InMotion, is a prospective randomized controlled trial where the study participants will be randomized to 12-weeks of physical training with creative movement as an intervention in addition to standard care (intervention group) or to standard care alone (control group). The target group consists of adults with SCZ or SCZ-similar condition.

The intervention consists of organized training sessions in group, 2 times a week. The control group receives standard medical care and gets access to the intervention in digital form after the study has ended. The outcomes are measured at baseline, after 6 and 12 weeks, 6 months and 12 months. At all follow-ups, data are collected for both the intervention and control groups. The trial is being conducted in Örebro, Sweden. The study follows the standard methodology of intervention research.

60 patients with SCZ will be recruited continuously by staff at the psychiatry at the university hospital in Örebro. When matched to inclusion and exclusion criteria, written and informed consent will be obtained from all participants willing to participate. 30 patients will be randomized to participate in creative physical training in addition to continuing their conventional treatment plan (SCZ-I group) and 30 patients will be randomized to control group and receive treatment as usual (SCZ-C). Randomization to SCZ-I and SCZ-C groups will be done by sealed envelopes given to the participants after baseline measures.

The intervention covers various themes through three different parts (4 weeks per part). The intervention was developed by a team consisting of physiotherapists, dance teachers, a neuroscientist and a psychiatrist, with the aim to improve clinical symptoms, physical fitness, cognitive skills and emotion regulations. The intervention is further described in Table 1. The exercise is partly accompanied with calm music and recorded nature sounds and partly made in silence listening to one's own bodily rhythm. The exercise consists of tasks related to cardio and strength training, balance, conscious breathing, body awareness, mental imagery (nature visualizations), flexibility, emotional expression, and movement anticipation together with the facilitator and fellow participants. All the tasks are practiced during a flow of 45- to 60-minute exercise without any major breaks. Complexity and physical intensity of the tasks will gradually increase over the 12-week intervention period.

The duration of the biweekly creative movement intervention will be from 45 minutes (week 1 and 2) to 60 minutes (week 3-12), the order and content of which is described in detail in Table 1. Throughout the intervention period, the participants will be encouraged to practice their favorite movements or relaxation techniques at home if they want to. The participants will get recordings of the sessions from the intervention coordinators in the research team, if they want to have support in practicing on their own at home. If a participant misses a session, they will get a text-message and an email with the video again, and encouragement to practice at home to keep up the frequency of two sessions a week, and the instructor will ask them if they have done so to ensure that it is important and relevant with regularity.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia diagnosis or schizophrenia similar condition, age 18-65 years, performing physical activity less than 150 min/week.

Exclusion Criteria:

* Current or recent history of substance abuse, bipolar disorder, severe autism, suicidal, severe physical illness, inability to read and understand the Swedish language and inability to interact with other people in a group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 45 minutes
  The Positive and Negative Syndrome Scale (PANSS) is an established psychiatric rating system that is an operationalized, drug-sensitive instrument that offers balanced representation of positive and negative symptoms and estimates their relationship to one another and to global (or general) psychopathology.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity scale (CGI-S) | 2.5 minutes
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
Clinical Global Impression - Improvement scale (CGI-I) | 2.5 minutes
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
The Calgary Depression Scale for Schizophrenics (CDSS) | 10 minutes
  The Calgary Depression Scale for Schizophrenia (CDSS) is a nine item clinician rated outcome measure that assesses the level of depression in people with schizophrenia.
Body Awareness Questionnaire (BAQ-sv) | 10 minutes
  Body Awareness Questionnaire includes 18 suggestions of four subgroups (changes in the body process, sleep-wake cycle, estimation of disease onset, and estimation of body reactions) and aims to determine the level of body awareness.
The personal and social performance scale (PSP) | 10 minutes
  The Personal Social Performance scale assesses socially useful activities, personal and social relationships, self-care and disturbing and aggressive behaviours.
EQ-5D-5L | 5 minutes
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Burden of Care - Visual Analogue Scale | 5 minutes
  Burden of Care is rated on a Visual Analogue Scale by a significant other, measuring the expressed burden in relation to the patient, the last month.
Physiological measures | 15 minutes
  Blood pressure measured by blood pressure monitor, resting heart rate, and breathing frequency
Body measures | 5 minutes
  Weight, length, BMI and waistline will be measured
Motion Capture | 60 minutes
  Movement of the participants will be recorded with the Qualisys Motion Capture device during the movement intervention
fNIRS, EEG, and eye-tracking | 45 minutes
  Cortical activity and eye movements will be measured from the patients with a combined EEG-fNIRS cap and eye-tracking glasses in stillness (baseline brain activity) and when doing conventional tasks measuring cognitive skills, emotion regulation and movement imitation
Postural stability test/balance | 10 minutes
  Measuring postural sway while person is standing on a forceplate
Chair stand test | 3 minutes
  Chair stand test to measure strength in the legs
Everyday activity | 7 days
  Everyday activity is measured by an accelerometer which the participants will carry with them for seven days in a row to collect the amount of time spent sedentary, and active, and the intensity of the activity
Blood samples | 5 minutes
  Blood samples including triglycerides, cholesterol, HDL, VLDL, HbA1, CRP, IL1b, IL6, TNFa, Hb, LPK, TPK, ASAT, ALAT, Natrium, Potassium and Creatinin
Interviews | 60 minutes
  Qualitative semistructured interviews with 15-20 persons after the intervention. Both participants and related parties get to share their experience of the intervention as well as eventual effects from it

CONTACTS AND LOCATIONS:
Overall Officials: Mats Eriksson, Professor, Principal Investigator — Örebro University, Sweden
Locations (2):
- Sweden (2):
  - Region Örebro county, Örebro
  - Örebro University, Örebro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poikonen H, Duberg A, Eriksson M, Eriksson-Crommert M, Lund M, Moller M, Msghina M. "InMotion"-Mixed physical exercise program with creative movement as an intervention for adults with schizophrenia: study protocol for a randomized controlled trial. Front Hum Neurosci. 2023 Jul 5;17:1192729. doi: 10.3389/fnhum.2023.1192729. eCollection 2023. PMID 37476005